CLINICAL TRIAL: NCT06604104
Title: Seeing Through Their Eyes - Towards Defining Visual Frailty in Ageing
Brief Title: Visual Frailty in Ageing
Acronym: VFiA
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC24002; REC reference: 24/SS/0021/AM01 (Other: South East Scotland Research Ethics Committee 01); IRAS project ID: 338463 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Frailty; Age-Related Macular Degeneration; Functional Status; Mental Health; Depression; Anxiety; Cognitive Impairment; Visual Impairment
Keywords: Visual frailty; Frailty; Ageing; Reading performance; Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Frailty; Macular Degeneration; Psychological Well-Being; Depression; Anxiety Disorders; Cognitive Dysfunction; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to define visual frailty and refine monitoring for an ageing population. It involves piloting a visual frailty assessment tool in a cohort of patients aged 60 and above with a known diagnosis of Age-related Macular Degeneration (AMD) in Princess Alexandra Eye Pavilion (PAEP), Anne Rowling Clinic which is hosting the NHS Low Visual Aid Clinic, or any other NHS Lothian facility treating patients with Age-related Macular Degeneration (AMD). The main questions it aims to answer are:

* What is visual frailty and how can it be assessed or predicted in the global ageing population using visual acuity, reading performance, functional status, mental health and systemic co-morbidities?
* What is the relationship between visual acuity, reading performance, ocular diagnosis, co-morbidities, mental health, and functional status?

Participants will have the following data collected from them from either Princess Alexandra Eye Pavilion, Anne Rowling Clinic which is hosting the NHS Low Visual Aid Clinic, or any other NHS Lothian facility treating patients with Age-related Macular Degeneration (AMD):

* Visual acuity (both distance and near)
* Reading performance
* Functional status
* Mental health
* Co-morbidities

Data will also be collected remotely (by phone call) from both the participants and their carers/relatives about their perceptions of visual frailty.

Expert opinion will be sought from optometrists and ophthalmologists about the concept of visual frailty using an online survey.

DETAILED DESCRIPTION:
This is a mixed methods observational cross-sectional study that will consist of designing a tool to measure visual frailty and piloting it in a cohort of participants in the ageing population. The study will be implemented over a period of three years: literature review to define visual frailty and designing of the tool in the first year, recruitment of participants and performing a pilot and a validation study in the second year and thesis write-up in the final year.

Participants aged 60 and above with a known diagnosis of advanced Age-related Macular Degeneration (AMD) will be recruited from Princess Alexandra Eye Pavilion (PAEP) macular clinic, Anne Rowling Clinic which is hosting the NHS Low Visual Aid Clinic, or any other NHS Lothian facility treating patients with Age-related Macular Degeneration (AMD).

The visual frailty index will consist of results from visual acuity, reading performance, functional status, mental health and co-morbidities. This tool will be piloted in a cohort of 20 patients with advanced AMD. The internal consistency of the tool will be determined at this phase of the project.

In addition to visual frailty, physical frailty will also be assessed in this cohort to enable analysis and establishment of the relationship between the two.

The patients with AMD and their relatives/carers will be invited to participate in remote data collection about their perspectives on visual frailty.

Best corrected distance and near visual acuity will be assessed and recorded. Reading performance will consist of reading speed and reading acuity which will be automatically measured using Digital Radner that will be acquired and installed before the implementation of the study.

Functional status will be assessed using Lawton and Brody Instrumental Activities of Daily Living (IADL) Scale.

Mental health will consist of depression, anxiety, and cognitive impairment that will be assessed using General Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), and Six-item Cognitive Impairment Test (6-CIT) respectively. All these are validated tools.

Physical frailty will be assessed using the FRAIL scale which relies on functions of fatigue, resistance, ambulation, illnesses and loss of weight.

Information about co-morbidities will be retrieved from the patients' health record through National Health Service (NHS) Lothian.

The data to be collected remotely from both the patients and their relatives/carers will be done through a phone call which will be scheduled during the hospital appointment. These calls will be recorded for analysis. They will then be transcribed verbatim, coded, and themes will be generated during the analysis.

In addition to defining and designing a tool to measure visual frailty, expert input will be sought from optometrists and ophthalmologists about this topic using an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be residents of Scotland aged 60 years and above with a known diagnosis of advanced AMD.
* The patients should be receiving treatment from Princess Alexandra Eye Pavilion (PAEP) for at least 6 months and should be responding positively to the treatment. This is to rule out poor results due to either not receiving medication or non-compliance.
* The participants should be able to provide informed consent before taking part in the study.

Exclusion Criteria:

* Participants who cannot speak and read English language will not be included in this pilot study. However, non-English speakers will be included in the future together with interpreters at the validation phase of the developed tool.
* Participants who have undergone invasive ocular surgery like cataract extraction in their previous visit.
* The potential participants who fail to provide or do not provide informed consent will not be included in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 60 and above with a known diagnosis of advanced Age-related Macular Degeneration (AMD) will be recruited from Princess Alexandra Eye Pavilion (PAEP) macular clinic.
  Their relatives or carers will also participate in the study but their data will be collected remotely. The term relatives/carers will be restricted to spouses/partners or children of the patients with advanced AMD.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Visual frailty | Within the first day of enrollment into the study.
  This will be assessed in units of visual frailty index. This is a pilot study and the visual frailty index will be derived from the results from the outcomes measures described below. These outcome measures include visual acuity, reading performance, functional status, mental health, and co-morbidities.

SECONDARY OUTCOMES:
Visual acuity | Within the first day of enrollment into the study.
  Visual acuity will be assessed using logMAR charts and will be recorded in logMAR units.
Reading performance | Within the first day of enrollment into the study.
  To be assessed using Digital Radner. The results will be recorded in terms of reading speed (measured in words per minute) and reading acuity (measured in logRAD)
Functional status | Within the first day of enrollment into the study.
  To be assessed using Lawton and Brody Instrumental Activities of Daily Living scale. The score on this scale ranges from 0 to 8 for women and 0 to 5 for men. The lower value (0) corresponds to low function or being dependent while the highest values (8 or 5) correspond to high function or being independent.
Mental health (Depression) | Within the first day of enrollment into the study.
  This will be assessed using Patient Health Questionnaire -9 tool. The scores are classified as: 1-4: Minimal depression; 5-9: Mild depression; 10-14: Moderate depression; 15-19: Moderately severe depression; and 20-27: Severe depression
Mental health (Anxiety) | Within the first day of enrollment into the study.
  This will be assessed using the Generalized Anxiety Disorder - 7 tool. The scores are classified as: 0-4: Minimal anxiety; 5-9: Mild anxiety; 10-14: Moderate anxiety; and 15-21: Severe anxiety
Mental health (Cognitive Impairment) | Within the first day of enrollment into the study.
  This will be assessed using the 6-item Cognitive Impairment Test. The score ranges from 0 to 28 in which 0-7 are considered normal and 8 or more are considered to be more significant.
Co-morbidities | Within the first day of enrollment into the study.
  These will be collected from the medical records of participants and a simple count of the conditions will be used.
Physical frailty | Within the first day of enrollment into the study.
  This will be assessed using the frail scale which relies on functions of fatigue, resistance, ambulation, illnesses and loss of weight. The scores range from 0 to 5. A score of 0 represents robust health status; 1-2 means participant is pre-frail; and 3-5 means the participant is Frail.
Correlation between visual frailty and physical frailty | This will be done immediately after assessment of both visual frailty and physical on the first day.
  Results of visual frailty and physical frailty will be analysed to establish the correlation between the two.
Correlation between Age-related macular degeneration and frailty | This will be done immediately after assessment of physical frailty on the first day.
  Age-related macular degeneration stage will be retrieved from the medical records and frailty will be assessed using the FRAIL scale which relies on functions of fatigue, resistance, ambulation, illnesses and loss of weight.
Perception about visual frailty | Within 4 weeks from the assessment date of visual frailty.
  This qualitative data will be remotely collected through a phone call from both the patients with AMD and their relatives/carers
Expert opinion about visual frailty | From enrolment to the end of the study, an average of approximately 3 months.
  This will be collected via an online survey from optometrists and ophthalmologists.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cackett, Principal Investigator — Princess Alexandra Eye Pavilion; Ian Underwood, Study Director — School of Engineering, University of Edinburgh
Locations (2):
- United Kingdom (2):
  - The Princess Alexandra Eye Pavilion, Edinburgh, Scotland
  - Anne Rowling Clinic, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data from the results section will be made available.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Rahi JS, Cumberland PM, Peckham CS. Visual impairment and vision-related quality of life in working-age adults: findings in the 1958 British birth cohort. Ophthalmology. 2009 Feb;116(2):270-4. doi: 10.1016/j.ophtha.2008.09.018. Epub 2008 Dec 16. PMID 19091416
- [Background] Polack S, Kuper H, Wadud Z, Fletcher A, Foster A. Quality of life and visual impairment from cataract in Satkhira district, Bangladesh. Br J Ophthalmol. 2008 Aug;92(8):1026-30. doi: 10.1136/bjo.2007.134791. PMID 18653592
- [Background] Peters D, Heijl A, Brenner L, Bengtsson B. Visual impairment and vision-related quality of life in the Early Manifest Glaucoma Trial after 20 years of follow-up. Acta Ophthalmol. 2015 Dec;93(8):745-52. doi: 10.1111/aos.12839. Epub 2015 Sep 18. PMID 26382936
- [Background] Dzenana RA, Smaila H. Quality of life of elderly people with visual impairment in relation to the degree of visual impairment. Human Research in Rehabilitation. 2022, DOI: 10.21554/hrr.042207
- [Background] Rahman MS, Rahman MA, Ali M, Rahman MS, Maniruzzaman M, Yeasmin MA, Ahmed NAMF, Abedin MM, Islam SMS. Determinants of depressive symptoms among older people in Bangladesh. J Affect Disord. 2020 Mar 1;264:157-162. doi: 10.1016/j.jad.2019.12.025. Epub 2019 Dec 16. PMID 32056745
- [Background] Dong X, Ng N. Contribution of multiple pathways to the relationship between visual impairment and depression: Explaining mental health inequalities among older Chinese adults. J Affect Disord. 2021 Jan 1;278:350-356. doi: 10.1016/j.jad.2020.09.068. Epub 2020 Sep 14. PMID 33002726
- [Background] Demmin DL, Silverstein SM. Visual Impairment and Mental Health: Unmet Needs and Treatment Options. Clin Ophthalmol. 2020 Dec 3;14:4229-4251. doi: 10.2147/OPTH.S258783. eCollection 2020. PMID 33299297
- [Background] Court H, McLean G, Guthrie B, Mercer SW, Smith DJ. Visual impairment is associated with physical and mental comorbidities in older adults: a cross-sectional study. BMC Med. 2014 Oct 17;12:181. doi: 10.1186/s12916-014-0181-7. PMID 25603915
- [Background] Itokazu M, Ishizaka M, Uchikawa Y, Takahashi Y, Niida T, Hirose T, Ito A, Yakabi A, Endo Y, Sawaya Y, Igawa T, Kobayashi K, Hara T, Watanabe M, Kubo A, Urano T. Relationship between Eye Frailty and Physical, Social, and Psychological/Cognitive Weaknesses among Community-Dwelling Older Adults in Japan. Int J Environ Res Public Health. 2022 Oct 11;19(20):13011. doi: 10.3390/ijerph192013011. PMID 36293591
- [Background] Klein BE, Klein R, Knudtson MD, Lee KE. Relationship of measures of frailty to visual function: the Beaver Dam Eye Study. Trans Am Ophthalmol Soc. 2003;101:191-6; discussion 196-9. PMID 14971577
- [Background] Klaver CC, Wolfs RC, Vingerling JR, Hofman A, de Jong PT. Age-specific prevalence and causes of blindness and visual impairment in an older population: the Rotterdam Study. Arch Ophthalmol. 1998 May;116(5):653-8. doi: 10.1001/archopht.116.5.653. PMID 9596502
- [Background] Wolfram C, Schuster AK, Elflein HM, Nickels S, Schulz A, Wild PS, Beutel ME, Blettner M, Munzel T, Lackner KJ, Pfeiffer N. The Prevalence of Visual Impairment in the Adult Population. Dtsch Arztebl Int. 2019 Apr 26;116(17):289-295. doi: 10.3238/arztebl.2019.0289. PMID 31196384
- [Background] Prince MJ, Wu F, Guo Y, Gutierrez Robledo LM, O'Donnell M, Sullivan R, Yusuf S. The burden of disease in older people and implications for health policy and practice. Lancet. 2015 Feb 7;385(9967):549-62. doi: 10.1016/S0140-6736(14)61347-7. Epub 2014 Nov 6. PMID 25468153
- [Background] Blindness in the elderly. Lancet. 2008 Oct 11;372(9646):1273. doi: 10.1016/S0140-6736(08)61527-5. No abstract available. PMID 18929885
- [Background] Salvi SM, Akhtar S, Currie Z. Ageing changes in the eye. Postgrad Med J. 2006 Sep;82(971):581-7. doi: 10.1136/pgmj.2005.040857. PMID 16954455
- [Background] Loh KY, Ogle J. Age related visual impairment in the elderly. Med J Malaysia. 2004 Oct;59(4):562-8, quiz 569. PMID 15779599
- [Background] Varadaraj V, Lee MJ, Tian J, Ramulu PY, Bandeen-Roche K, Swenor BK. Near Vision Impairment and Frailty: Evidence of an Association. Am J Ophthalmol. 2019 Dec;208:234-241. doi: 10.1016/j.ajo.2019.08.009. Epub 2019 Aug 26. PMID 31465753
- [Background] Partridge L, Deelen J, Slagboom PE. Facing up to the global challenges of ageing. Nature. 2018 Sep;561(7721):45-56. doi: 10.1038/s41586-018-0457-8. Epub 2018 Sep 5. PMID 30185958
- [Background] Restrepo HE, Rozental M. The social impact of aging populations: some major issues. Soc Sci Med. 1994 Nov;39(9):1323-38. doi: 10.1016/0277-9536(94)90364-6. PMID 7801169
- [Background] Shrestha LB. Population aging in developing countries. Health Aff (Millwood). 2000 May-Jun;19(3):204-12. doi: 10.1377/hlthaff.19.3.204. PMID 10812800
- See also: Ageing published by The United Nations — https://www.un.org/en/global-issues/ageing#:~:text=Globally%2C%20the%20population%20aged%2065%20and%20over%20is,Northern%20America%20could%20be%20aged%2065%20or%20over.
- See also: WHO- Blindness and vision impairment — https://www.who.int/news-room/fact-sheets/detail/blindness-and-visual-impairment
- See also: Eye frailty Awareness by the Japan Ophthalmology Society — https://www.eye-frail.jp/